CLINICAL TRIAL: NCT00757770
Title: Study to Assess the Clinical Consistency of Three Production Lots of GSK Biologicals' HRV Vaccine in Terms of Immunogenicity and Safety When Given to Healthy Infants at 2 and 4 Months of Age
Brief Title: Assessment of Clinical Consistency of Three Production Lots of GSK Biologicals' HRV Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 444563/033
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Rotavirus
Keywords: Gastroenteritis
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group HRV Lot A (Experimental)
  Interventions: Biological: Rotarix
- Group HRV Lot B (Experimental)
  Interventions: Biological: Rotarix
- Group HRV Lot C (Experimental)
  Interventions: Biological: Rotarix
- Group Placebo (Active Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rotarix — Two oral doses.
  Arms: Group HRV Lot A; Group HRV Lot B; Group HRV Lot C
Biological: Placebo — Two oral doses; The placebo consist of all components of the study vaccine i.e. excipients and buffer, but no RV particles.
  Arms: Group Placebo

SUMMARY:
The purpose of this study is to evaluate the lot-to-lot consistency of three production lots of GSK Biologicals' HRV vaccine in terms of immunogenicity and safety in healthy infants aged 2 months at the time of first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Child is unlikely to remain in the study area for the duration of the study.
* Previous confirmed occurrence of rotavirus gastroenteritis.
* Gastroenteritis within 7 days preceding the study vaccine administration.
* Household contact with an immunosuppressed individual or pregnant woman.
* Use of antibiotics during the period starting from 7 days before dose 1 of vaccine(s).
* Planned administration of a vaccine (other than routine pediatric vaccines) not foreseen by the study protocol during the period starting from 14 days before each dose of study vaccine(s) and ending 14 days after.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal tract or other serious medical condition as determined by the investigator.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* Acute disease at time of enrollment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 854 (Actual)
Dates: Start 2003-08; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Serum anti-rotavirus Immunoglobulin A (IgA) antibody concentration expressed as Geometric Mean Concentrations (GMCs). | Two months after Dose 2.

SECONDARY OUTCOMES:
Serum anti-rotavirus IgA antibody concentration expressed as GMCs in a subset of subjects. | Two months after Dose 1.
Seroconversion rates to anti-rotavirus IgA antibody | Two months after Dose 1 (in a subset of subjects) and Dose 2 (all subjects).
Vaccine take rates in a subset of subjects. | Two months after each dose
Presence of rotavirus in stool samples in a subset of subjects | On the day of each vaccination and on planned days following each vaccination.
For each type of solicited symptom, occurrence of the symptom | During the 8-day follow-up period after each vaccine dose
Occurrence of unsolicited symptoms | During the 31-day follow-up period after each vaccine dose.
Occurrence of serious adverse events | Throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Cali Colombia, Colombia
- GSK Investigational Site, Mexico City, Mexico
- GSK Investigational Site, Lima, Peru
- GSK Investigational Site

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Lopez P, Herrera JFG, Cervantes Y, et al. Three consecutive production lots of the human monovalent RIX4414 G1P(8) rotavirus vaccine, Rotarix™ induce a consistent immune response in Latin American infants. Proc 4th World Congress Pediatr Infect Dis, Warsaw, Poland, 2005.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 444563/033 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 444563/033 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 444563/033 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 444563/033 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 444563/033 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 444563/033 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register